CLINICAL TRIAL: NCT04652154
Title: Transitioning Young Patients' Health Care Trajectories (TpT) Bridging the Gap Between Mental and Somatic Health Services "Tjenester på Tvers"
Brief Title: Transitioning Young Patients' Health Care Trajectories
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/344
Record Dates: First submitted 2020-10-31; First posted 2020-12-03 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-02

CONDITIONS: Health Care Utilization; Mental Health Impairment; Child, Only; Multi-morbidity
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Participants are invited to either intervention or treatment as usual
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Control group is recieving treatment as ususal
  Interventions: Other: Transitioning young patients' health care trajectories
- Intervention group (Experimental): The intervention group getting the new assessment by a complementary professional team
  Interventions: Other: Transitioning young patients' health care trajectories

INTERVENTIONS:
Other: Transitioning young patients' health care trajectories — New intervention where the patient with multi-referrals to specialist health service meet with a complementary professional team consisting of doctor, psychologist and physioterapist aiming clarify the child's condition through shared decison-making and agreeing upon treatment plans for the child

SUMMARY:
The project aims to transition the approach used to care for children with complex conditions and care pathways into a more holistic and coordinated model. The traditional model where specialists independently treat single diseases, makes joint and coordinated decisions about patients with multiple and unclear conditions difficult. In particular there is a gap between mental and somatic services.

In preparation for re-designing the care model, several pre-studies are conducted, both a register study and a collection of user reported experiences. Built on the results, we have invented multi-disciplinary teams of complementary competences including paediatricians, psychologists, and physiotherapists to meet the patient and family. The study includes:

* To implement the new team intervention in a clinical case-control study
* To scientifically evaluate the intervention
* To systematise lessons learned in regard to potential spread across systems and patient groups Children 6-16 years together with family and professionals will constitute the team. The assessment aims to clarify the patient's condition through shared decision making and to develop a treatment plan for the child. It is a clinical randomised controlled trial where TpT children will be compared to children following treatment as usual. It includes a one year follow-up regarding a set of evaluation domains: provider perspectives, user-centred experiences and outcomes, as well as health care outcomes.

DETAILED DESCRIPTION:
200 children with multi-referrals will be invited to either intervention or treatment as usual at their third or more referral to Haukeland university hospital.

In the intervention group the child and family will meet a complementary team of professionals for more than two hours aimimg to get a clarification of the patient's condition and giving coping strategies for their condition. Outcome defined as better mental health and quality of life as well as increased school attendence are some of the measures being collected. These outcomes will be compared to the control group after 12 mth.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-16 years,
* Previous referred to specialist health care service for 3 or more times, including mental health service as well paediatric service.

Exclusion Criteria:

* Not within age range
* Less than 3 referrals

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Contentment with the intervention - Patient | Through study completion, an average of 2 years
  Patient evaluate the intervention - A questionnaire for the study has been developed "Contentment of the TpT intervention (Patient)" with two items and for each item has a score 1-4 and 4 is most positive.
Contentment with the intervention - Parents | Baseline
  Parents evaluate the intervention - A questionnaire for the study has been developed "Contentment of the TpT intervention (Parent)" with two items and score for each item has 1-4 and 4 is most positive.
Contentment with the intervention - Parents | Through study completion, an average of 2 years
  Parents evaluate the intervention - A questionnaire for the study has been developed "Contentment of the TpT intervention (Parent)" with two items and score for each item has 1-4 and 4 is most positive.
Contentment with the intervention - Professionals | Through study completion, an average of 2 years
  Professionals evaluate the intervention - A questionnaire for the study has been developed Usefulness of the TpT intervention with two items and score for each item has 1-4 and 4 is most positive.
Mental health status | Baseline
  Strenght and Difficulty Questionnaire (SDQ) is a mental health screening questionnaire. It constitutes 20 items, with five items in each of the four subscales:emotional problems, hyperactivity/inattention, conduct problems, and peer problems.
Mental health status | 1 year after the intervention
  Strenght and Difficulty Questionnaire (SDQ) is a mental health screening questionnaire. It constitutes 20 items, with five items in each of the four subscales:emotional problems, hyperactivity/inattention, conduct problems, and peer problems.
Mental health status | 2 year after the intervention
  Strenght and Difficulty Questionnaire (SDQ) is a mental health screening questionnaire. It constitutes 20 items, with five items in each of the four subscales:emotional problems, hyperactivity/inattention, conduct problems, and peer problems.
Quality of Life: KIDSCREEN-27 Barne/ungdomsversjon 8-18år | Baseline
  Using KIDSCREEN-27 to evaluate Quality of Life, caregiver provide information in five dimensions these are Rasch scales: Physical Well-Being (5 items), Psychological Well-Being (7 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items).
  Each item has a scale of five where 1 is "not at all" is worse outcome and 5 "very much" is the best outcome.
Quality of Life: KIDSCREEN-10 Barne/ungdomsversjon 8-18år | 1 year after the intervention
  Using KIDSCREEN-10 to evaluate Quality of Life, caregiver provide information in five dimensions these are Rasch scales: Physical Well-Being (5 items), Psychological Well-Being (7 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items).
  Each item has a scale of five where 1 is "not at all" is worse outcome and 5 "very much" is the best outcome.

SECONDARY OUTCOMES:
Contact with specialist healthcare | 1 year after the intervention after the intervention
  Post evaluation of use of health services - numbers of new referrals

CONTACTS AND LOCATIONS:
Overall Officials: Hans Olav Instefjord, Master, Study Chair — Haukeland University Hospital
Locations (1):
- Haukeland universitet sykehus, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elgen I, Lygre RB, Arli A, Heggestad T. An interdisciplinary intervention for children with complex health complaints; a feasibility study of selection criteria. Front Pediatr. 2023 Sep 14;11:1167528. doi: 10.3389/fped.2023.1167528. eCollection 2023. PMID 37780046
- [Result] Elgen I, Heggestad T, Tronstad R, Greve G. Bridging the Gap for Children With Compound Health Challenges: An Intervention Protocol. Front Pediatr. 2021 Dec 22;9:721926. doi: 10.3389/fped.2021.721926. eCollection 2021. PMID 35004532
- [Result] Heggestad T, Greve G, Skilbrei B, Elgen I. Complex care pathways for children with multiple referrals demonstrated in a retrospective population-based study. Acta Paediatr. 2020 Dec;109(12):2641-2647. doi: 10.1111/apa.15250. Epub 2020 Apr 17. PMID 32159873
- [Result] Elgen I, Lygre R, Greve G, Griffiths S, Heggestad T. Interdisciplinary Approaches Suggested for Children With Multiple Hospital Referrals Presenting With Non-specific Conditions. Front Pediatr. 2021 Apr 7;9:656939. doi: 10.3389/fped.2021.656939. eCollection 2021. PMID 33898364
- [Result] Lygre RB, Gjestad R, Norekval TM, Mercer SW, Elgen IB. An interdisciplinary intervention for children and adolescents with multiple referrals and complex health complaints: a feasibility study. BMC Health Serv Res. 2023 Nov 11;23(1):1241. doi: 10.1186/s12913-023-10250-y. PMID 37951903
- [Result] Lygre RB, Thuen VM, Gjestad R, Norekval TM, Greve G, Mildestvedt T, Elgen IB. How can we improve specialist health services for children with multi-referrals? Parent reported experience. BMC Health Serv Res. 2020 Aug 24;20(1):786. doi: 10.1186/s12913-020-05666-9. PMID 32831078